CLINICAL TRIAL: NCT05243394
Title: Evaluating the Effects of a Treadmill Gait Training Protocol in a Gamified Virtual Reality Environment With tDCS in Parkinson's Disease: Randomized Controlled Trial
Brief Title: Effects of a Treadmill Gait Training Protocol in a Gamified Virtual Reality Environment With tDCS in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat de Lleida (Other)
Collaborators: University of Turku (Other); University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Helena Fernández-Lago, Lecturer, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI20/00403
Record Dates: First submitted 2022-01-20; First posted 2022-02-17 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Parkinson Disease
Keywords: Virtual Reality; Gamification; tDCS; Treadmill gait training; Dual Task
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: 3 groups of 22 participants will each follow a different treatment option.
Who Masked: Outcomes Assessor
Masking Description: The outcome measuring assessors will not know from which group any of the participants comes from, and will have no interaction with any of the interventions applied.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gamified virtual reality environtment + tDCS + treadmill gait training (Experimental): The first group will follow an 18-session gait training protocol for 6 weeks. Duration of the sessions will progressively increase from 20 to 45 minutes from first session to last. They will be immersed in a gamified virtual reality environment in which they will interact with the in-game ambient by having their feet represented on the screen and move as their own on the treadmill. They will also receive tDCS for the first 20 minutes of each session.
  Interventions: Other: Gamified virtual reality treadmill gait training with tDCS
- Gamified virtual reality environtment + treadmill gait training (Experimental): The second group will follow an 18-session gait training protocol for 6 weeks. Duration of the sessions will progressively increase from 20 to 45 minutes from first session to last. They will be immersed in a gamified virtual reality environment in which they will interact with the in-game ambient by having their feet represented on the screen and move as their own on the treadmill.
  Interventions: Other: Gamified virtual reality treadmill gait training
- Treadmill gait training (Active Comparator): The third group will follow an 18-session gait training protocol for 6 weeks. Duration of the sessions will progressively increase from 20 to 45 minutes from first session to last.
  Interventions: Other: Treadmill gait training

INTERVENTIONS:
Other: Gamified virtual reality treadmill gait training with tDCS — Progressive treadmill gait training in a gamified virtual reality environment with tDCS
  Arms: Gamified virtual reality environtment + tDCS + treadmill gait training
Other: Gamified virtual reality treadmill gait training — Progressive treadmill gait training in a gamified virtual reality environment
  Arms: Gamified virtual reality environtment + treadmill gait training
Other: Treadmill gait training — Progressive treadmill gait training
  Arms: Treadmill gait training

SUMMARY:
The study aims to compare the effects of treadmill gait training in a gamified virtual reality environment with tDCS versus treadmill gait training in a gamified virtual reality environment versus treadmill training in people with Parkinson's Disease.

DETAILED DESCRIPTION:
Treadmill gait training has been stablished as a solid gait rehabilitation option for people with Parkinson's Disease. However, gait training by itself fails to address the cognitive aspect needed for safe walking, which could be affected by situations in which concurrent tasks must be managed simultaneously to gait. It also lacks motivational aspects key to keep people with Parkinson's Disease adhered to treatment. Virtual reality and gamification are posed as useful tools to address both these issues, turning training into a more engaging activity and allowing complicated gait situations to be trained in a safe environment. Transcranial direct current stimulation (tDCS) could be combined with these mentioned treatment options, which could reinforce the learning of motor and cognitive skills during training.

The aim of this study is to evaluate the effects of the inclusion of a gamified virtual reality environment to a treadmill gait training program with tDCS in PD compared to the same training protocol with virtual reality and without it

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease
* Stage II - III in the Hoehn and Yahr Scale during ON state
* Ability to walk for 10 minutes independently without stop

Exclusion Criteria:

* Significant cognitive decline based on mini mental status examination (MMSE <23)
* Severe auditory or visual deficits
* Other neurological/psychiatric conditions
* Any kind of cardiovascular complications that contraindicates physical activity
* Clinical history of any brain surgery or deep brain stimulation device

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Stride lenght | 14 weeks
  Stride length will be recorded while walking on a 10-meter aisle with an inertial sensor system while the patient is asked to walk at preferred, very slow, slow, medium, high and very high speed. Will be measured in meters (m).
Speed | 14 weeks
  Speed will be recorded while walking on a 10-meter aisle with an inertial sensor system while the patient is asked to walk at preferred, very slow, slow, medium, high and very high speed. Will be measured in meters per second (m/s).
Step cadence | 14 weeks
  Step cadence will be recorded while walking on a 10-meter aisle with an inertial sensor system while the patient is asked to walk at preferred, very slow, slow, medium, high and very high speed. Will be measured in Hertz (Hz).
Stride Length during Dual Task | 14 weeks
  Stride length will be recorded while walking on a 10-meter aisle with an inertial sensor system while listening to an audio recording, in which patients will hear certain set words and will have to remember how many times they are mentioned (Phoneme Monitoring Paradigm Dual Task). Participants will be asked to walk at preferred speed. Will be measured in meters (m).
Speed during Dual Task | 14 weeks
  Speed will be recorded while walking on a 10-meter aisle with an inertial sensor system while listening to an audio recording, in which patients will hear certain set words and will have to remember how many times they are mentioned (Phoneme Monitoring Paradigm Dual Task). Participants will be asked to walk at preferred speed. Will be measured in meters per second (m/s).
Step cadence during Dual Task | 14 weeks
  Step cadence will be recorded while walking on a 10-meter aisle with an inertial sensor system while listening to an audio recording, in which patients will hear certain set words and will have to remember how many times they are mentioned (Phoneme Monitoring Paradigm Dual Task). Participants will be asked to walk at preferred speed. Will be measured in Hertz (Hz).
Stride Length Variation Coeficient | 14 weeks
  Based on standard deviation and mean values of Stride Length data, a new variable will be calculated to assess the variability of stride length in participants' gait. Formula will be the following: (Standard deviation/mean Stride Length)100
Stride Length Variation Coeficient during Dual Task | 14 weeks
  Based on standard deviation and mean values of Stride Length data, a new variable will be calculated to assess the variability of stride length in participants' gait. Formula will be the following (data from Dual Task variable): (Standard deviation/mean Stride Length)100
Step Cadence Variation Coeficient | 14 weeks
  Based on standard deviation and mean values of step cadence data during Dual Task, a new variable will be calculated to assess the variability of step cadence in participants' gait. Formula will be the following: (Standard deviation/mean Step Cadence)100
Step Cadence Variation Coeficient during Dual Task | 14 weeks
  Based on standard deviation and mean values of step cadence data during Dual Task, a new variable will be calculated to assess the variability of step cadence in participants' gait. Formula will be the following (data from Dual Task variable): (Standard deviation/mean Step Cadence)100

SECONDARY OUTCOMES:
Total Cognitive Performance | 14 weeks
  A battery of executive function tests will be applied, which in combination will allow for a total cognitive performance calculation. The used tests to calculate the Total Cognitive Performance are: Trail Making Test, Digit Span Backwards, Word Fluency Phonemic and Semantic, Wisconsin Card Sorting Test, Corsi Block Test, and Tower of London Test. These test scores will be converted to z-test scores and integrated with a formula to obtain the Total Cognitive Performance score.
Unified Parkinson's Disease Rating Scale (UPDRS) | 14 weeks
  The UPDRS is made up of 42 items grouped into four subscales: Section I-mentation, behavior and mood; Section II-activities of daily living (scored for "on" and "off"); Section III-motor exam; and Section IV-complications. Items from Sections I to III are scored on a 4-point scale. Section IV contains dichotomous items and items scored on a 4-point scale for duration or severity. Higher scores indicate more severe impairment.
Hoehn & Yahr | 14 weeks
  Assess symptom progression in Parkinson's Disease based on a 5-stage scale, in which stage 1 is the most autonomous and stage 5 implies bedridden or wheelchair-bound patients unless assisted.
Parkinson's Disease Questionnaire 39 | 14 weeks
  Patient-reported 39 item questionnaire to assess Parkinson's Disease related quality of life and health status across 8 dimensions of daily living. Higher scores indicate worse quality of life.
MiniBest Test | 14 weeks
  14-item test to assess dynamic balance. Lower scores mean a worse balance condition.
Montreal Cognitive Assessment | 14 weeks
  30-question test to assess cognitive function. Lower scored mean a worse cognitive status.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Fernández-Lago, Principal Investigator — Universitat de Lleida
Locations (1):
- Institut de Recerca Biomèdica de Lleida, Lleida, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yogev-Seligmann G, Hausdorff JM, Giladi N. The role of executive function and attention in gait. Mov Disord. 2008 Feb 15;23(3):329-42; quiz 472. doi: 10.1002/mds.21720. PMID 18058946
- [Background] Shahed J, Jankovic J. Motor symptoms in Parkinson's disease. Handb Clin Neurol. 2007;83:329-42. doi: 10.1016/S0072-9752(07)83013-2. No abstract available. PMID 18808920
- [Background] Mehrholz J, Kugler J, Storch A, Pohl M, Hirsch K, Elsner B. Treadmill training for patients with Parkinson Disease. An abridged version of a Cochrane Review. Eur J Phys Rehabil Med. 2016 Oct;52(5):704-713. Epub 2016 Mar 4. PMID 26940123
- [Background] Dockx K, Bekkers EM, Van den Bergh V, Ginis P, Rochester L, Hausdorff JM, Mirelman A, Nieuwboer A. Virtual reality for rehabilitation in Parkinson's disease. Cochrane Database Syst Rev. 2016 Dec 21;12(12):CD010760. doi: 10.1002/14651858.CD010760.pub2. PMID 28000926
- [Background] Schootemeijer S, van der Kolk NM, Ellis T, Mirelman A, Nieuwboer A, Nieuwhof F, Schwarzschild MA, de Vries NM, Bloem BR. Barriers and Motivators to Engage in Exercise for Persons with Parkinson's Disease. J Parkinsons Dis. 2020;10(4):1293-1299. doi: 10.3233/JPD-202247. PMID 32925106
- [Background] Broeder S, Nackaerts E, Heremans E, Vervoort G, Meesen R, Verheyden G, Nieuwboer A. Transcranial direct current stimulation in Parkinson's disease: Neurophysiological mechanisms and behavioral effects. Neurosci Biobehav Rev. 2015 Oct;57:105-17. doi: 10.1016/j.neubiorev.2015.08.010. Epub 2015 Aug 20. PMID 26297812
- [Background] Mirelman A, Rochester L, Reelick M, Nieuwhof F, Pelosin E, Abbruzzese G, Dockx K, Nieuwboer A, Hausdorff JM. V-TIME: a treadmill training program augmented by virtual reality to decrease fall risk in older adults: study design of a randomized controlled trial. BMC Neurol. 2013 Feb 6;13:15. doi: 10.1186/1471-2377-13-15. PMID 23388087
- [Derived] Bosch-Barcelo P, Climent-Sanz C, Martinez-Navarro O, Masbernat-Almenara M, Pakarinen A, Ghosh PK, Fernandez-Lago H. A treadmill training program in a gamified virtual reality environment combined with transcranial direct current stimulation in Parkinson's Disease: Study protocol for a randomized controlled trial. PLoS One. 2024 Jul 16;19(7):e0307304. doi: 10.1371/journal.pone.0307304. eCollection 2024. PMID 39012877
- [Derived] Bosch-Barcelo P, Masbernat-Almenara M, Martinez-Navarro O, Tersa-Miralles C, Pakarinen A, Fernandez-Lago H. A gamified virtual environment intervention for gait rehabilitation in Parkinson's Disease: co-creation and feasibility study. J Neuroeng Rehabil. 2024 Jun 24;21(1):107. doi: 10.1186/s12984-024-01399-6. PMID 38915103